CLINICAL TRIAL: NCT06219447
Title: Innovative Models for Taking on and Tele-rehabilitation of Neuropsychomotor and Language Skills in Children and Adolescents With Congenital and Acquired Developmental Disabilities (TABLET-TOSCANA).
Brief Title: Tele-rehabilitation in Subjects With Congenital and Acquired Developmental Disabilities
Acronym: TABLETOSCANA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Giovanni Cioni (Other)
Collaborators: Azienda USL Toscana Nord Ovest (Other); Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor-Investigator, Giovanni Cioni, MD, PhD, IRCCS Fondazione Stella Maris
Organization: IRCCS Fondazione Stella Maris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TABLET-TOSCANA
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Congenital and Acquired Developmental Disabilities
Keywords: Information and Communication Technologies; Tele-rehabilitation; Neuropsychomotor skills; Language skills; Neurodevelopmental disabilities; Organizational models; Feasibility

STUDY DESIGN:
Intervention Model Description: It will be a waitlist study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Children will be immediately trained through the TABLET TOSCANA technologies (VRRS Home Tablet or Medico Amico Kids APP) for a cycle of 3 months.
  Interventions: Device: VRRS Home Tablet or Medico Amico Kids APP
- Waitlist group (No Intervention): Children will continue standard care for 3 months and after that they will be guaranteed to be enrolled for the next 3-month cycle through the TABLET TOSCANA technologies (VRRS Home Tablet or Medico Amico Kids APP).

INTERVENTIONS:
Device: VRRS Home Tablet or Medico Amico Kids APP — Tele-rehabilitation (TR) permits intensive and personalized intervention monitored by clinicians in an ecological friendly, home setting. The VRRS Home Kit, comprising a tablet and peripheral devices, permits TR of cognitive, speech and motor functions. These peripherals such as sensors and balances allow motor rehabilitation across different body districts involved (upper and lower limbs, trunk). Touch screen activities, enables neuropsychological and speech therapy sessions. Medico Amico APP, offers a wide library of cognitive, language and motor exercises, stratified by difficulty levels, targeting specific functions. An avatar guides real-time movements, offering visual references. Adjustable parameters include duration, repetitions, difficulty, speed, movement amplitude. Both technologies facilitate TR sessions via a dedicated platform, that can occur in real-time, involving interaction with patients, or independently with continuous monitoring by clinical staff.
  Arms: Experimental group

SUMMARY:
The COVID-19 emergency has led to the complete closure of all rehabilitation services, both public and/or private, across Italy, including the region of Tuscany. Among the various consequences of the COVID-19 pandemic, a significant negative indirect impact on children with neurodevelopmental disabilities and their families was observed. Specifically within Tuscany, a substantial decline occurred in rehabilitative interventions, including physiotherapy, language therapy, and neuropsychological therapy. Despite these challenges, some healthcare facilities responded by initiating tele-rehabilitation treatments, even if on a limited scale, following the recommendations of scientific societies within the field. In this framework, TABLET-TOSCANA project has been developed, with the overall aim of developing innovative organizational models to ensure the continuity of care for treatment and tele-rehabilitation of neuro-psychomotor and language functions in children with congenital and acquired developmental disabilities. The present proposal aims to evaluate the feasibility of this approach and the economic sustainability of employing the implemented technologies to promote tele-rehabilitation as possible territorial care taking. Additionally, the study aims to conduct a preliminary efficacy evaluation by analyzing pre-post treatment changes identified in outcome measures, providing valuable insights into the potential benefits of this tele-rehabilitation proposal.

DETAILED DESCRIPTION:
Tele-rehabilitation is designed as a timely, intensive, and personalized intervention aimed to provide access to rehabilitation services monitoring by the clinical staff. This intervention enables activities to be carried out in an ecological and home-based environment, following the key components of evidence-based neuropsychological and motor rehabilitation. Different studies, including those conducted in Italy, have demonstrated promising results through the application of Information and Communication Technologies (ICTs) in rehabilitation, even in the developmental age. Tele-rehabilitation, therefore, could be particularly suitable to support the treatment of children with neurodevelopmental disorders and their families, in order to enable continuity of care by extending rehabilitation programs into home settings, fostering family involvement, continuous monitoring by the clinical team. This was even more relevant during the critical period of the COVID-19 emergency, as the use of ICT proved indispensable for the uninterrupted care of patients and their families and, consequently, mitigate the adverse consequences of care disruptions on the short-, medium-, and long-term neuropsychological outcomes, stress levels, and overall quality of life for the entire family.

The overarching aim of the TABLET-TOSCANA project is to develop innovative organizational models that foster the continuity of care and tele-rehabilitation for neuro-psychomotor and language functions in children with congenital and acquired developmental disabilities. Throughout the project, two technologies currently employed in the cognitive, motor, and speech rehabilitation of adult patients will be adapted for the pediatric population: (i) the VRRS Home Tablet and (ii) the Medico Amico Kids APP. Later, these technologies will be tested in the pediatric and young adult populations through a waitlist-type randomized pilot study evaluating usability, acceptability and economic sustainability by the principal stakeholders (patients, their caregivers and all members of the multidisciplinary clinical team, such as child neuropsychiatrists, physiatrists, neuropsychologists, developmental neuropsychomotricity therapists, physical therapists, speech therapists). This project unfolds into three main phases.

(i) The initial phase involves the implementation of the Medico Amico Kids APP and the VRRS Home Tablet in order to adapt them to the pediatric population's specific needs. Specifically, both technologies will facilitate professionals in monitoring, conducting teleconsultations, and delivering treatment programs through online or offline tele-rehabilitation sessions. The clinical team, in relation to their expertise, will meticulously analyze the library of motor, cognitive and language exercises currently available in both systems in order to implement it in collaboration with Khymeia bioengineers to enhance usability for the pediatric population.

(ii) The middle phase will focus on technology validation: 100 subjects (80 children and 20 young adults) will be recruited in a pilot study. It will be a waitlist study to ensure that all enrolled patients will be eligible for the experimental treatment. Subjects will be selected and stratified according to diagnosis (congenital or acquired developmental disorder group), functional gross-motor level (GMFCS I-II/GMFCS III-IV), age (6-10/11-15/16-20/21-30), type of organizational model, and technology (APP vs. Home Tablet). After the evaluation, participants will be randomly assigned to either the experimental group (EG) (providing a 3-month tele-rehabilitation) or the waitlist group (WG) (continuing traditional rehabilitation care for the same duration). All children will be evaluated before and after 3 months of intervention with standardized clinical tests. At the end of tele-rehabilitation of EG, ad-hoc questionnaires, aligned with standardized tools and investigation criteria from a literature review, will be administered to assess feasibility and sustainability across various areas, including usability and acceptability, defined by ISO/DIS 9241-11 standard and the Technology Acceptance Model, respectively.

(iii) During the final phase both feasibility and the preliminary efficacy data will be processed. In particular, feasibility data will comprise not only the ad-hoc designed questionnaire but also parameters such as: study and rehabilitation adherence, number of drop out, number of sessions completed within the period of treatment defined, encountered technical problems hindering tele-rehabilitation execution, and acceptance evaluations. Regarding the efficacy data, given the heterogeneity of the clinical population in terms of both chronological age and functional profile, a wide set of tests with normative data covering an extended age range has been selected for the assessment of cognitive, neuropsychological, motor, and language abilities. This approach will allow for the selection of the tests most suited to each patient's functional profile. Furthermore, treatment effectiveness will be examined using the Goal Attainment Scale (GAS), a rehabilitation outcome measure, which is scored based on individual goals hypothesized and achieved throughout the intervention. Finally, the merging of these datasets will contribute to the formulation of innovative organizational models, incorporating tele-assistance and tele-rehabilitation pathways.

ELIGIBILITY:
Inclusion Criteria:

* Congenital or acquired developmental disabilities;
* Ages from 6 to 30 years old at the time of recruitment;
* Cognitive functioning that allows sufficient understanding of proposed activities and cooperation in exercises, investigated by appropriate rating scales (WPPSI-III or WPPSI-IV or WISC-IV or WAIS-IV or LEITER-R or LEITER-3 or RAVEN Matrices).
* Sufficient distance from the clinical center to allow periodic in-person assessment of progress
* Possibility to have internet access at home
* Caregivers able to be committed to and cooperate in an intensive rehabilitation home-based program.
* Manual Ability Classification System (MACS) level < V

Exclusion Criteria:

* Severe comorbidities and/or severe cognitive disability
* MACS level V

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2024-02-12 (Estimated); Study Completion 2024-06-12 (Estimated)

PRIMARY OUTCOMES:
Tele-rehabilitation feasibility measures: Study adherence | T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)
  Rate of acceptance of the participation in the study calculated as the number of eligible participants that agree to join the project.
Tele-rehabilitation feasibility measures: Adherence to training | T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)
  Total number of training sessions completed on the total number of sessions scheduled by the clinicians, expressed as a ratio.
Tele-rehabilitation feasibility measures: Number of dropouts | T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)
  Number of participants that will not complete the all study procedures.
Tele-rehabilitation feasibility measures: Number of sessions completed in the target time | T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)
  Total number of training session completed in the timeframe setted by clinicians.
Tele-rehabilitation feasibility measures: Technical problems encountered that prevent the program from running | T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)
  Number of issues and malfunctioning experimented by clinicians and families during the training sessions.
Feasibility questionnaire | T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)
  In order to investigate the feasibility of the system used and the compliance of children, their families and the clinicians, will be carried out an ad hoc questionnaire at the end of the training, during the post-intevention assessment. The answer questionnaire is built with a 5-point likert scale; higher scores means a greater feasibility for the stakeholder who filled the questionnaire.

SECONDARY OUTCOMES:
Changes in Sustained attention subtest of Leiter 3 | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  Sustained Attention is a subtest of the Leiter-3 non-verbal cognitive scale. It allows the assessment of visual sustained attention through barrage tasks of increasing complexity within a set time frame. The number of correctly selected target elements are recorded. Raw scores range from 0 to 217, while standardized score range from 0 to 20. Higher scores revealed better performances.
Changes in visual attention CP subtest of Italian Battery for ADHD (BIA) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  CP is a subtest of the Italian battery for ADHD (BIA). This subtest allows the assessment of visual sustained attention through barrage tasks of increasing complexity. Number of omissions are recorded (ranging from 0 to 54), and then converted in percentile scores. Lower raw scores reveal better performances.
Changes in Conners' Parent Rating Scale - Brief version | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  Conner's Parent Rating Scale is a parent report questionnaire about clinical behaviours in children, with a specific focus on ADHD symptoms. Parents have to rate each item administered according to the how often this behaviour is shown by their child in the last month, circling the best option on a 3-point Likert scale. Four indices are then extracted and converted in T scores: oppositional behaviour (scores range 0 to 18), inattention/cognitive problems (scores range 0 to 18), hyperactivity (scores range 0 to 18), ADHD index (scores range 0 to 36). Higher scores reveal clinical behaviour.
Changes in Visuo-motor precision subtest of NEPSY II | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  Visuo-motor precision is a subtest of the NEPSY II battery, used for the assessment of the ability to follow a narrow path with the pencil in an accurate and quick way. Total execution time and number of errors are recorded and then converted in percentile or standardized scores (ranging from 1 to 19). Higher scores reveal a better performance.
Changes in Developmental Test Of Visuo-Motor Integration | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  Visuo-motor integration task is a paper and pencil test requiring geometrical figures to be copied, assessing difficulties in integrating or coordinating visual perceptual and motor (finger and hand movement) abilities. The number of figures correctly reproduced is recorded and then converted in standardized scores. Raw scores range from 0 to 27. Higher scores reveal a better performance.
Changes in digit span forwards and backward subtests of BVN | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  Digit span is a subtest of BVN battery both for children aged 5-11 and for 12-18 years old, allowing the assessment of short term and working memory abilities in the verbal domain though the repetition of a sequence of numbers of increasing length, following the same or a reverse order. The length of the last sequence correctly retrieved is recorded as the span, ranging from 3 to 9 in the forward condition and from 2 to 8 in the backward. Higher span reveals better performance.
Changes in Corsi Block Tapping test subtest of BVS-Corsi | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  Corsi Block Tapping task Is a subtest of the Italian BVS-Corsi battery, assessing short term and working memory abilities in the verbal domain though the repetition of a sequence (of increasing length) of blocks tapped by examiners, following the same or a reverse order.
  The length of the last sequence correctly retrieved is recorded as the span, ranging from 3 to 8 in the forward condition and from 2 to 7 in the backward. Higher span reveals better performance.
Changes in Behaviour Rating inventory of executive function (BRIEF 2/P) for parents | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  Questionnaire administered to parents in order to assess executive functioning in daily life contexts. Parents have to rate each item administered according to the how often this behaviour is shown by their child in the last six months, circling the best option on a 3-point Likert scale. In the BRIEF 2 version, 9 scales are then extracted and converted in T scores: inhibition (ranging 8-24), self-monitoring (ranging 4-12), shift (ranging 8-24), emotional regulation (ranging 8-24), initiate (ranging 5-15), working memory (ranging 8-24), plan/organize (ranging 8-24), task monitoring (ranging 5-15), material organization (ranging 6-18); in the BRIEF P version, 5 scales are then extracted and converted in T scores: inhibition (ranging 16-48), shift (ranging 10-30), emotional regulation (ranging 10-30), working memory (ranging 17-51), plan/organize (ranging 10-30). Composite scores could be also calculated. Higher scores reveal clinical behaviours.
Changes in route finding subtest of NEPSY II | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  Route finding is a subtest of the NEPSY II battery, assessing the ability to use a small schematic map to locate a target on a larger schematic map, therefore orienting in visuo-spatial coordinates. Raw scores range from 0 to 10, and then percentile scores are extracted. Higher scores reveal a better performance.
Changes in arrow subtest of NEPSY II | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  Arrow subtest of the NEPSY II battery, assess the ability to judge lines orientation, considering and estimating direction, in distance, orientation and angularity. Raw scores range from 0 to 38, and then percentile scores are extracted. Higher scores reveal a better performance.
Changes in reading and writing tasks of Dyslexia and Developmental Dysortography Evaluation-2 (DDE-2) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This battery evaluates reading and writing skills in children. In this study will be assess two subtests: Test 2 and 3 (reading words and non-words), Test 6 and 7 (writing words and non-words under dictation).
Changes in reading and writing tasks of Martini Battery | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This battery evaluates reading and writing skills in children. The subtests including activities of reading and writing flat bisyllabic and trysillabic words, bisyllabic and trysillabic words with consonantal group.
Changes in writing tasks of Battery for the assessment of writing and orthographic competence-2 (BVSCO-2) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  The BVSCO-2 is a comprehensive tool for assessing all aspects involved in writing's learning process: handwriting, orthographic competence and production of written text. This battery is for children attending primary and secondary school (6-14). In this study will be assessed two subtests: text writing under dictation and spontaneous text writing based on figure stories.
Changes in reading and text comprehension of MT Battery- Third Version (MT-3) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This battery assess reading and text comprehension skills, identify reading difficulties and make a diagnosis of dyslexia in primary and secondary school (6-14 years old).
Changes in lexical comprehension of Peabody Picture Vocabulary Test - Revised (PPVT-R) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This is a receptive vocabulary test for children aged 3.9 to 11.6 years that uses nouns, verbs and adjectives of increasing difficulty as stimulus words for a total of 175 tables. The raw score is the number of correct responses in the critical range, then Lexical Quotient (LQ) can be calculated, it's an age-equivalent standard score.
Changes in Children's Grammatical Comprehension Test (TCGB) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This is a multiple-choice figurative test that assesses grammatical comprehension in children aged 3.6 to 8 years. The test consists of 76 sentences, which refer to 8 main types of grammatical structures.
Changes in Gross Motor Function Measure 88 (GMFM-88) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  The GMFM-88 assess gross motor function in children between 5 months to 16 years of age according to five dimensions: (i) Lying and Rolling, (ii) Sitting, (iii) Crawling and Kneeling, (iv) Standing, and (v) Walking, Running and Jumping. There is a four-point ordinal scoring system for each GMFM item. Then, the item scores can be summed in order to calculate raw and percentage scores for each of the five dimensions, the selected target areas, and the total GMFM-88 score. The higher the score, the better the gross motor skills.
Changes in 6 minutes walking test (6MWT) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  The 6MWT assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. it can be used in preschool children (2-5 years), children (6-12 years) adults (18-64 years), elderly adults (65+) with a wide range of diagnoses including. An increase in the distance walked during 6 minute indicates improvement in basic mobility.
Changes in Pediatric Balance Scale (PBS) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  The PBS is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children with mild to moderate motor impairments. The scale consists of 14 items criterion-references that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Changes in Functional Reach Test (FRT) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  It is a functional assessment tool of dynamic balance evaluated in one simple task in standing position. It measures the maximum distance an individual can reach with an anterior shift with a fixed base of support. Scores are determined by assessing the difference between the start and end position is the reach distance (measured in inches or cm). Greater value (distance) = better balance and decreased falls risk. Three trials are done and average of last two noted.
Changes in Timed Up and Go (TUG) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  The TUG test assesses mobility, balance, walking ability, and fall risk. It is a functional dynamic balance test which measures the time it takes for the patient to stand up from a chair, walk 3 meters, turn around, walk back, and sit down.
Changes in the Assisting Hand Assessment (AHA) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This assessment measures the assisting hand performance in children with unilateral upper limb disabilities, during bimanual performances. It can be used for children aged between 18 months and 18 years, with playful session made of semi-structured activities calibrated on the different ages (different board games). Is a standardized criterion-referenced test and the sum of scores may vary between 20 and 80, where a higher score indicates a higher ability level; the scaled score ranges between 0 and 100 and is a transformation of the sum score to a percentage distribuition within the scale, where 100 indicates that all test items were performed with the highest scores, and 0 means that all test items were performed with the lowest points.
Changes in Both Hand Assessment (BoHA) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This assessment measures both hands performance in children with bilateral cerebral palsy, during bimanual performances. It can be used for children aged between 18 months and 12 years, with playful session made of semi-structured activities calibrated on the different ages (different board games). Is a standardized criterion-referenced test and the sum of scores may vary between 20 and 80, where a higher score indicates a higher ability level; the scaled score ranges between 0 and 100 and is a transformation of the sum score to a percentage distribuition within the scale, where 100 indicates that all test items were performed with the highest scores, and 0 means that all test items were performed with the lowest points.
Changes in Melbourne Assessment 2 (MA2) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  It is a valid and reliable criterion-referenced test that measures unilateral upper extremity quality of movement in children, aged 2.5 to 15 years, with neurological impairments according four elements: (i) Range of movement, (ii) Accuracy of reach and placement, (iii) Dexterity of grasp, release and manipulation and (iv) Fluency of movement. Scoring is completed across the 30 score items using a three-, four- or five-point scale and individually defined scoring criteria. Item scores relating to each element of movement measured are summed within the corresponding sub-scale. A child's final score on the MA2 is reported as four separate scores, one for each element of movement quality measured. A higher score indicates a higher upper limb ability investigated.
Changes in Box and Block Test (BBT) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  It measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations from childhood to adults. The score is given by the number of blocks carried from one compartment to the other in one minute. Higher scores on the test indicate better gross manual dexterity. The two hands will be both tested starting from the dominant one.
Changes in Movement Disorders - Childhood Rating Scale Revised (MD-CRS R) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  The MD-CRS R is a standardized and validated, child-oriented rating scale aimed at describing and assessing movement disorders in children and adolescents aged 4-18 years, and their influence on activities of daily living or motor function in different regions of the body at rest and while performing specific tasks. All items are rated on a five-point ordinal scale (0-4), in which the lowest score means better performance.
Changes in Test of Visual Perception and Visuo-motor Integration (TPV) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  TPV is a test for the evaluation of visuo-perceptual and visuo-motor integration skills. In the study the investigators will assess the subtests: (i) Copying/reproduction subtest: the child sees figures that he have to copy; (ii) Visual/motor speed: the child is asked to draw distinctive designs inside the target figures; (iii) hand-eye coordination: the child is asked to draw some lines inside bands of different widths; (iv) spatial relationship: the child is asked to connect some dots to reproduce the target figure.
Changes in Abilhand Kids | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This questionnaire measures the manual abilities of children with CP (6-15 years old), with a particular reference to the independence in achieving some goals of everyday life, exploring if some activities are easily performed, if they present some difficulties or if they are impossible. It can be answered by parents or children and it requires 10 minutes.
Changes in Movement Assessment Battery for Children- Second Edition (MABC-2) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This battery evaluates movement difficulties in 3 to 16 years children and adolescents. The tasks are divided by age range and organised into three sections: manual dexterity, aiming and catching and balance. Scores are provided in standard scores and percentiles and are interpreted by using a traffic light system: green light (scores above 15◦ percentile), meaning typical motor performances; yellow light (scores between 5◦ and 15◦ percentile), indicating a risk for motor impairment; red light (scores below 5◦ percentile), identifying a significant motor function impairment.
Changes in Praxic and Motor Coordination Skills-2nd Edition (APCM-2) | T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)
  This test aims to assess motor and praxis skills in children aged between 2-8 years, with age group-specific performance tests. APCM-2 allows early detection of motor-praxic coordination deficit, and the scores make it possible to detail the functional profile of each case, obtained by calculating the distance from the normative mean and referring to percentile values (5°, 10°, 25°), in order to identify for each scale the specific functions, both the most integral and the most impaired.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No